CLINICAL TRIAL: NCT04243343
Title: A Randomized, Controlled, Multi-site Trial of a Specific Acupuncture Protocol for the Treatment of Plantar Fasciosis
Brief Title: Specific Acupuncture Protocol for the Treatment of Plantar Fasciosis
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: brett rasmussen (U.S. Federal Agency)
Responsible Party: Sponsor-Investigator, brett rasmussen, Principal Investigator, Mike O'Callaghan Military Hospital
Organization: Mike O'Callaghan Military Hospital (U.S. Federal Agency)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: FWH20200060H
Record Dates: First submitted 2020-01-22; First posted 2020-01-28 (Actual); Last update posted 2022-01-28 (Actual); Status verified 2022-01

CONDITIONS: Plantar Fascitis
Keywords: Plantar fasciosis; acupuncture; electrostimulation; primary care
MeSH Terms: interventions — Methods; Standard of Care

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Intervention + Standard of care (Experimental): Acupuncture with electrostimulation plus standard of care prescribed home exercise program.
  Interventions: Device: Intervention + Standard of care
- Standard of care (Active Comparator): Standard of care prescribed home exercise program.
  Interventions: Other: Standard of care

INTERVENTIONS:
Device: Intervention + Standard of care — Acupuncture with electrostimulation plus standard of care prescribed home exercise program for treatment of plantar fasciosis.
  Arms: Intervention + Standard of care
Other: Standard of care — Standard of care prescribed home exercise program for treatment of plantar fasciosis.
  Arms: Standard of care

SUMMARY:
Determine if the addition of a specific acupuncture protocol to a standard of care prescribed exercise program is more effective at improving pain and function in adult patients with plantar fasciosis.

DETAILED DESCRIPTION:
This is a randomized, controlled, multi-site trial investigating whether a specific acupuncture protocol can improve pain and function in adults with plantar fasciosis when added to standard of care treatment. The investigators hypothesize that there will be a significant improvement in both pain and functional outcomes, both acutely and over time, in the experimental group compared to the control group.

ELIGIBILITY:
**Patients must be able to get care at Nellis Air Force Base, Scott Air Force Base, or Eglin Air Force Base (a military installation) in order to participate in this study**

Inclusion Criteria:

* Male and female DoD beneficiaries, aged 18 to 74 years, who have been diagnosed with plantar fasciosis (in one or both of their feet) OR
* Patients meeting criteria of pain in the bottom of the foot/heel with first steps in the morning & tender to palpation over the medial calcaneal tubercle (where the plantar fascia inserts).

Those with acute and chronic diagnoses will be included.

Exclusion Criteria:

* Pregnant
* Any of the following in the foot being included into the study:

  * Active cellulitis of lower extremity
  * Prior surgery for plantar fasciosis
  * Steroid injections in the last 12 weeks for plantar fasciosis; if received in last 12 weeks subjects will be offered to be involved in the study after they have completed a 12 -week wash out period.
  * If they have every had any prior acupuncture for plantar fasciosis using the defined Deep Ankle Local Periosteal points, any regenerative therapy to include proliferation therapy or platelet rich plasma therapy in the last 12 weeks for plantar fasciosis; if received in last 12 weeks subject will be offered to be involved in the study after they have completed a 12-week wash out period.
  * Botox injections for plantar fasciosis injections in the last 12 weeks for plantar fasciosis; if received in last 12 weeks subject will be offered to be involved in the study after they have completed.

Ages: 18 Years to 74 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 72 (Actual)
Dates: Start 2020-06-01 (Actual); Primary Completion 2021-11-02 (Actual); Study Completion 2021-11-02 (Actual)

PRIMARY OUTCOMES:
Defense and Veterans Pain Rating Scale (DVPRS) | visit 1 (Day 1)
  The DVPRS consists of an 11-point numerical rating scale with 0 indicating no pain and 10 indicating severe pain. It has been confirmed for reliability and validity in measuring both acute and chronic pain, and is currently the standard for pain measurement throughout DoD and VA health systems. The DVPRS has demonstrated linear scale qualities allowing parametric methods to be used
Defense and Veterans Pain Rating Scale (DVPRS) | visit 2 (week 2)
  The DVPRS consists of an 11-point numerical rating scale with 0 indicating no pain and 10 indicating severe pain. It has been confirmed for reliability and validity in measuring both acute and chronic pain, and is currently the standard for pain measurement throughout DoD and VA health systems. The DVPRS has demonstrated linear scale qualities allowing parametric methods to be used
Defense and Veterans Pain Rating Scale (DVPRS) | visit 3 (week 4)
  The DVPRS consists of an 11-point numerical rating scale with 0 indicating no pain and 10 indicating severe pain. It has been confirmed for reliability and validity in measuring both acute and chronic pain, and is currently the standard for pain measurement throughout DoD and VA health systems. The DVPRS has demonstrated linear scale qualities allowing parametric methods to be used
Defense and Veterans Pain Rating Scale (DVPRS) | visit 4 (week 6)
  The DVPRS consists of an 11-point numerical rating scale with 0 indicating no pain and 10 indicating severe pain. It has been confirmed for reliability and validity in measuring both acute and chronic pain, and is currently the standard for pain measurement throughout DoD and VA health systems. The DVPRS has demonstrated linear scale qualities allowing parametric methods to be used
Defense and Veterans Pain Rating Scale (DVPRS) | visit 5 (week 12)
  The DVPRS consists of an 11-point numerical rating scale with 0 indicating no pain and 10 indicating severe pain. It has been confirmed for reliability and validity in measuring both acute and chronic pain, and is currently the standard for pain measurement throughout DoD and VA health systems. The DVPRS has demonstrated linear scale qualities allowing parametric methods to be used
Defense and Veterans Pain Rating Scale Supplemental Questions | visit 1 (Day 1)
  The DVPRS consists of an 11-point numerical rating scale with 0 indicating no pain and 10 indicating severe pain. For clinicians to evaluate the biopsychosocial impact of pain.
Defense and Veterans Pain Rating Scale Supplemental Questions | visit 2 (week 2)
  The DVPRS consists of an 11-point numerical rating scale with 0 indicating no pain and 10 indicating severe pain. For clinicians to evaluate the biopsychosocial impact of pain.
Defense and Veterans Pain Rating Scale Supplemental Questions | visit 3 (week 4)
  The DVPRS consists of an 11-point numerical rating scale with 0 indicating no pain and 10 indicating severe pain. For clinicians to evaluate the biopsychosocial impact of pain.
Defense and Veterans Pain Rating Scale Supplemental Questions | visit 4 (week 6)
  The DVPRS consists of an 11-point numerical rating scale with 0 indicating no pain and 10 indicating severe pain. For clinicians to evaluate the biopsychosocial impact of pain.
Defense and Veterans Pain Rating Scale Supplemental Questions | The DVPRS consists of an 11-point numerical rating scale with 0 indicating no pain and 10 indicating severe pain. visit 5 (week 12)
  For clinicians to evaluate the biopsychosocial impact of pain.
Foot function index revised short (FFI-R short) | visit 1 (Day 1)
  FFI-R short uses a likert questionnaire to document foot pain severity, foot stiffness, difficulty performing activities, activity limitation, and social issues related to affected foot.
  It consists of 23 self-reported items divided into 3 subcategories on the basis of patient values: pain, disability and activity limitation.The patient has to score each question on a scale from 0 (no pain or difficulty) to 10 (worst pain imaginable or so difficult it requires help), that best describes their foot over the past week.
Foot function index revised short (FFI-R short) | visit 2 (week 2)
  FFI-R short uses a likert questionnaire to document foot pain severity, foot stiffness, difficulty performing activities, activity limitation, and social issues related to affected foot.
  It consists of 23 self-reported items divided into 3 subcategories on the basis of patient values: pain, disability and activity limitation.The patient has to score each question on a scale from 0 (no pain or difficulty) to 10 (worst pain imaginable or so difficult it requires help), that best describes their foot over the past week.
Foot function index revised short (FFI-R short) | visit 3 (week 4)
  FFI-R short uses a likert questionnaire to document foot pain severity, foot stiffness, difficulty performing activities, activity limitation, and social issues related to affected foot.
  It consists of 23 self-reported items divided into 3 subcategories on the basis of patient values: pain, disability and activity limitation.The patient has to score each question on a scale from 0 (no pain or difficulty) to 10 (worst pain imaginable or so difficult it requires help), that best describes their foot over the past week.
Foot function index revised short (FFI-R short) | visit 4 (week 6)
  FFI-R short uses a likert questionnaire to document foot pain severity, foot stiffness, difficulty performing activities, activity limitation, and social issues related to affected foot.
  It consists of 23 self-reported items divided into 3 subcategories on the basis of patient values: pain, disability and activity limitation.The patient has to score each question on a scale from 0 (no pain or difficulty) to 10 (worst pain imaginable or so difficult it requires help), that best describes their foot over the past week.
Foot function index revised short (FFI-R short) | visit 5 (week 12)
  FFI-R short uses a likert questionnaire to document foot pain severity, foot stiffness, difficulty performing activities, activity limitation, and social issues related to affected foot.
  It consists of 23 self-reported items divided into 3 subcategories on the basis of patient values: pain, disability and activity limitation.The patient has to score each question on a scale from 0 (no pain or difficulty) to 10 (worst pain imaginable or so difficult it requires help), that best describes their foot over the past week.

CONTACTS AND LOCATIONS:
Overall Officials: Paul F Crawford, MD, Study Director — United States Air Force
Locations (3):
- United States (3):
  - 96th Medical Group, Eglin Air Force Base, Florida
  - Scott AFB, Belleville, Illinois
  - Mike O'Callaghan Military Medical Center, Nellis Air Force Base, Nevada

IPD SHARING:
Plan to Share IPD: No
We do not plan on sharing data

REFERENCES:
- [Background] Cotchett MP, Landorf KB, Munteanu SE. Effectiveness of dry needling and injections of myofascial trigger points associated with plantar heel pain: a systematic review. J Foot Ankle Res. 2010 Sep 1;3:18. doi: 10.1186/1757-1146-3-18. PMID 20807448
- [Background] Covey CJ, Mulder MD. Plantar fasciitis: How best to treat? J Fam Pract. 2013 Sep;62(9):466-71. PMID 24080555
- [Background] Glickman-Simon R, Wallace J. Acupuncture for knee osteoarthritis, chasteberry for premenstrual syndrome, probiotics for irritable bowel syndrome, yoga for hypertension, and trigger point dry needling for plantar fasciitis. Explore (NY). 2015 Mar-Apr;11(2):157-61. doi: 10.1016/j.explore.2014.12.009. Epub 2014 Dec 29. No abstract available. PMID 25682385
- [Background] Goff JD, Crawford R. Diagnosis and treatment of plantar fasciitis. Am Fam Physician. 2011 Sep 15;84(6):676-82. PMID 21916393
- [Background] Kumnerddee W, Pattapong N. Efficacy of electro-acupuncture in chronic plantar fasciitis: a randomized controlled trial. Am J Chin Med. 2012;40(6):1167-76. doi: 10.1142/S0192415X12500863. PMID 23227789
- [Background] Landorf KB, Twyford GN, Cotchett MP, Whittaker GA. Revised minimal important difference values for the visual analogue scale and Foot Health Status Questionnaire when used for plantar heel pain. J Foot Ankle Res. 2024 Dec;17(4):e70021. doi: 10.1002/jfa2.70021. PMID 39682003
- [Background] Li S, Shen T, Liang Y, Zhang Y, Bai B. Miniscalpel-Needle versus Steroid Injection for Plantar Fasciitis: A Randomized Controlled Trial with a 12-Month Follow-Up. Evid Based Complement Alternat Med. 2014;2014:164714. doi: 10.1155/2014/164714. Epub 2014 Jul 8. PMID 25114704
- [Background] Schwartz O, Levinson T, Astman N, Haim L. Attrition due to orthopedic reasons during combat training: rates, types of injuries, and comparison between infantry and noninfantry units. Mil Med. 2014 Aug;179(8):897-900. doi: 10.7205/MILMED-D-13-00567. PMID 25102533
- [Background] Owens BD, Wolf JM, Seelig AD, Jacobson IG, Boyko EJ, Smith B, Ryan MA, Gackstetter GD, Smith TC; Millennium Cohort Study Team. Risk Factors for Lower Extremity Tendinopathies in Military Personnel. Orthop J Sports Med. 2013 Jun 11;1(1):2325967113492707. doi: 10.1177/2325967113492707. eCollection 2013 Jan-Jun. PMID 26535232
- [Background] Roy TC. Diagnoses and mechanisms of musculoskeletal injuries in an infantry brigade combat team deployed to Afghanistan evaluated by the brigade physical therapist. Mil Med. 2011 Aug;176(8):903-8. doi: 10.7205/milmed-d-11-00006. PMID 21882780
- [Background] Scher DL, Belmont PJ Jr, Bear R, Mountcastle SB, Orr JD, Owens BD. The incidence of plantar fasciitis in the United States military. J Bone Joint Surg Am. 2009 Dec;91(12):2867-72. doi: 10.2106/JBJS.I.00257. PMID 19952249
- [Background] Thiagarajah AG. How effective is acupuncture for reducing pain due to plantar fasciitis? Singapore Med J. 2017 Feb;58(2):92-97. doi: 10.11622/smedj.2016143. Epub 2016 Aug 16. PMID 27526703
- [Background] Woitzik E, Jacobs C, Wong JJ, Cote P, Shearer HM, Randhawa K, Sutton D, Southerst D, Varatharajan S, Brison RJ, Yu H, van der Velde G, Stern PJ, Taylor-Vaisey A, Stupar M, Mior S, Carroll LJ. The effectiveness of exercise on recovery and clinical outcomes of soft tissue injuries of the leg, ankle, and foot: A systematic review by the Ontario Protocol for Traffic Injury Management (OPTIMa) Collaboration. Man Ther. 2015 Oct;20(5):633-45. doi: 10.1016/j.math.2015.03.012. Epub 2015 Mar 28. PMID 25892707
- [Background] Zhang SP, Yip TP, Li QS. Acupuncture treatment for plantar fasciitis: a randomized controlled trial with six months follow-up. Evid Based Complement Alternat Med. 2011;2011:154108. doi: 10.1093/ecam/nep186. Epub 2011 Feb 15. PMID 19933769
- [Background] Polomano RC, Galloway KT, Kent ML, Brandon-Edwards H, Kwon KN, Morales C, Buckenmaier C' 3rd. Psychometric Testing of the Defense and Veterans Pain Rating Scale (DVPRS): A New Pain Scale for Military Population. Pain Med. 2016 Aug;17(8):1505-19. doi: 10.1093/pm/pnw105. Epub 2016 Jun 6. PMID 27272528
- [Background] Nassif TH, Hull A, Holliday SB, Sullivan P, Sandbrink F. Concurrent Validity of the Defense and Veterans Pain Rating Scale in VA Outpatients. Pain Med. 2015 Nov;16(11):2152-61. doi: 10.1111/pme.12866. Epub 2015 Aug 8. PMID 26257151
- [Background] Faul F, Erdfelder E, Lang AG, Buchner A. G*Power 3: a flexible statistical power analysis program for the social, behavioral, and biomedical sciences. Behav Res Methods. 2007 May;39(2):175-91. doi: 10.3758/bf03193146. PMID 17695343
- [Background] Sloman R, Wruble AW, Rosen G, Rom M. Determination of clinically meaningful levels of pain reduction in patients experiencing acute postoperative pain. Pain Manag Nurs. 2006 Dec;7(4):153-8. doi: 10.1016/j.pmn.2006.09.001. PMID 17145489
- [Background] Holm, S. 1979. A simple sequential rejective multiple test procedure. Scand. J. Statistics, 6: 65-70.
- [Background] R Core Team. R: A language and environment for statistical computing. R Foundation for Statistical Computing, Vienna, Austria. 2016 URL http://www.R-project.org/.
- See also: General Hospital and Personal Use Therapeutic Devices — http://www.accessdata.fda.gov/scripts/cdrh/cfdocs/cfcfr/cfrsearch.cfm?fr=880.5580

DOCUMENTS (1):
  • Informed Consent Form (2021-02-23): https://cdn.clinicaltrials.gov/large-docs/43/NCT04243343/ICF_000.pdf